CLINICAL TRIAL: NCT00064363
Title: A Phase II Trial Of Talampanel In Patients With Recurrent High-Grade Gliomas
Brief Title: Talampanel in Treating Patients With Recurrent High-Grade Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 030207; 03-C-0207; CDR0000315425; NCT00061685 (obsolete NCT alias)
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult anaplastic astrocytoma; adult glioblastoma; adult anaplastic oligodendroglioma; adult mixed glioma; adult giant cell glioblastoma; adult gliosarcoma; adult brain stem glioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Astrocytoma; Glioblastoma; Oligodendroglioma; Glioma; Gliosarcoma | interventions — talampanel

INTERVENTIONS:
Drug: talampanel

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as talampanel use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This phase II trial is studying how well talampanel works in treating patients with recurrent, progressive high-grade glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of talampanel, in terms of 6-month progression-free survival, in patients with recurrent high-grade gliomas.
* Determine, preliminarily, the toxic effects of this drug in these patients.
* Determine, preliminarily, the quality of life of patients treated with this drug.
* Determine the pharmacokinetics of this drug in patients who are and who are not receiving enzyme-inducing antiepileptic drugs.

OUTLINE: Patients are stratified according to type of glioma (anaplastic astrocytoma vs glioblastoma multiforme). Patients in each stratum are assigned to 1 of 3 treatment groups according to concurrent enzyme-inducing antiepileptic drug use (yes, no, or valproic acid).

Patients in each group receive different doses of oral talampanel 3 times daily on days 1-42. Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, every 3 weeks during the first course, every 6 weeks before all subsequent courses, and then within 2 weeks of study completion.

Patients are followed within 2 weeks.

PROJECTED ACCRUAL: A total of 91 patients (50 with anaplastic astrocytoma and 41 with glioblastoma multiforme) will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed high-grade glioma, including any of the following:

  * Glioblastoma multiforme
  * Anaplastic astrocytoma
  * Anaplastic oligodendroglioma
  * Anaplastic mixed oligoastrocytoma
  * Malignant astrocytoma not otherwise specified

    * Patients with clinical and radiographic diagnosis of brain stem glioma are also eligible
* Evidence of tumor progression by MRI or CT scan

  * Scan must be performed while patient is on a stable steroid dose for at least 5 days
* Must have failed prior radiotherapy
* Residual disease after prior resection of recurrent or progressive tumor is allowed

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* More than 8 weeks

Hematopoietic

* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count at least 100,000/mm^3 (transfusion independent)
* Hemoglobin at least 10 g/dL (transfusion allowed)

Hepatic

* Bilirubin less than 2 times upper limit of normal (ULN)
* SGOT less than 2 times ULN
* No significant active hepatic disease

Renal

* Creatinine less than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min
* No significant active renal disease

Cardiac

* No significant active cardiac disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 effective methods of contraception during and for 2 months after study participation
* Able to swallow whole capsules
* No active infection requiring IV antibiotics
* No significant active psychiatric disease that would preclude use of the study drug
* No other significant uncontrolled medical illness that would preclude study participation
* No other active life-threatening malignancy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 1 week since prior interferon or thalidomide
* No concurrent anticancer immunotherapy

Chemotherapy

* At least 2 weeks since prior vincristine
* At least 3 weeks since prior procarbazine
* At least 6 weeks since prior nitrosoureas
* No other concurrent anticancer chemotherapy

Endocrine therapy

* See Disease Characteristics
* At least 1 week since prior tamoxifen
* Concurrent steroids for the control of increased intracranial pressure allowed

Radiotherapy

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy
* No concurrent anticancer radiotherapy

Surgery

* See Disease Characteristics
* Prior recent resection of recurrent or progressive disease allowed

Other

* Recovered from all prior therapy
* At least 1 week since prior noncytotoxic agents (e.g., isotretinoin), except for radiosensitizers
* At least 4 weeks since prior investigational agents
* At least 4 weeks since prior cytotoxic therapy
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-06; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Progression at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Howard A. Fine, MD, Study Chair — NCI - Neuro-Oncology Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States

REFERENCES:
- [Result] Iwamoto FM, Kreisl TN, Kim L, Duic JP, Butman JA, Albert PS, Fine HA. Phase 2 trial of talampanel, a glutamate receptor inhibitor, for adults with recurrent malignant gliomas. Cancer. 2010 Apr 1;116(7):1776-82. doi: 10.1002/cncr.24957. PMID 20143438